CLINICAL TRIAL: NCT04076319
Title: Implementing CAPABLE in Permanent Supportive Housing
Brief Title: Implementing CAPABLE in PSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Benjamin F. Henwood, Associate Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UP-19-00361
Record Dates: First submitted 2019-08-27; First posted 2019-09-03 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Accidental Fall; Frailty; Depression; Activities of Daily Living; Housing Problems
MeSH Terms: conditions — Frailty; Depression | interventions — elderberry extract

STUDY DESIGN:
Intervention Model Description: Waitlist control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPABLE (Other): CAPABLE Intervention
  Interventions: Behavioral: CAPABLE: Community Aging in Place-Advancing Better Living for Elders

INTERVENTIONS:
Behavioral: CAPABLE: Community Aging in Place-Advancing Better Living for Elders — CAPABLE is a client-directed home-based intervention that consists of time-limited services from an occupational therapist, a nurse, and a handyman working collaboratively with the older adult client. In most cases, the OT makes 6 visits, the RN makes 4 visits, and a handyman makes 1 to 2 visits to make any modifications to a person's home during a 6-month period. The first visits for the OT and RN are usually 90 minutes each and the later ones are usually an hour each. Visits are spaced to enable older adults to practice new strategies learned in the previous visit. There should be a clear "conclusion/graduation," with the older adult understanding how to use their new skills and apply them to future situations.

SUMMARY:
This pilot project seeks to implement an intervention known as CAPABLE (Community Aging in Place-Advancing Better Living for Elders) for formerly homeless adults living in permanent supportive housing. This home-based intervention that consists of time-limited services (no more than 6-months) from an occupational therapist, a nurse, and a handyman is intended to improve functioning and decrease falls among this population that prematurely ages and is at increased fall risk.

DETAILED DESCRIPTION:
Permanent supportive housing (PSH) using a housing first approach is an evidence-based intervention to end chronic homelessness by providing low-barrier affordable housing paired with flexible health and social services. In Los Angeles County (LAC), where the number of PSH units is expected to increase dramatically over the next 10 years, clinical guidelines and/or standards for support services are lacking. This is especially problematic given the that the target population is older and prematurely aging. The chronically homeless population in the United States has an average age approaching 60 years old and experiences accelerated aging, including an elevated prevalence of geriatric syndromes such as functional impairment, falls, and urinary incontinence that can jeopardize PSH tenants' ability to live independently and age in place. Current support services are not equipped to address these needs, which ultimately jeopardizes the success of PSH to maintain high rates of housing stability while tenants "age in place."

The investigators propose conducting a pilot project to implement the CAPABLE model in PSH. CAPABLE, which stands for "Community Aging in Place-Advancing Better Living for Elders" is a client-directed home-based intervention that consists of time-limited services (no more than 6-months) from an occupational therapist, a nurse, and a handyman working collaboratively with the older adult client. CAPABLE was developed to target older adults who are returning to independent living after hospitalization and has been shown to improve functioning (activities of daily living - ADLs and instrumental activities of daily living - IADLs), decrease falls and nursing home admissions, and reduce healthcare costs based on multiple studies including several randomized control trials. CAPABLE has the potential to be used in PSH as a model of support services that can address needs of prematurely aging tenants, which could help transform PSH from an intervention that ends homeless to an intervention that addresses homelessness and supports successful aging in place.

The specific aims of this study are to:

1. Examine the impact of CAPABLE on PSH client outcomes (e.g. ADLs, IADLs, falls). This aim will be accomplished using a pre-/post-design with a wait-list control group.
2. Determine what adaptations, if any, need to be made to implement CAPABLE in PSH. The investigators will accomplish this aim using the Dynamic Adaptation Process (DAP) implementation approach, which was designed to allow for an evidenced-based practice to be adapted in a planned and considered, rather than ad hoc, manner.

Important to note is that this project was conducted during the COVID-19 pandemic so that adaptations to CAPABLE may be due to the context of the pandemic as opposed to being implemented in PSH.

ELIGIBILITY:
Inclusion Criteria:

* Older than 50 years in age
* cognitively intact or have only mild cognitive impairment
* have some or a lot of difficulty performing ADLs
* tenant of Skid Row Housing Trust

Exclusion Criteria:

* see above

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin F Henwood, PhD, Principal Investigator — University of Southern California
Locations (1):
- Skid Row Housing Trust, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate CAPABLE: CAPABLE is a client-directed home-based intervention that consists of time-limited services from an occupational therapist, a nurse, and a handyman working collaboratively with the older adult client. In most cases, the OT makes 6 visits, the RN makes 4 visits, and a handyman makes 1 to 2 visits to make any modifications to a person's home during a 6-month period. The first visits for the OT and RN are usually 90 minutes each and the later ones are usually an hour each. Visits are spaced to enable older adults to practice new strategies learned in the previous visit. There should be a clear "conclusion/graduation," with the older adult understanding how to use their new skills and apply them to future situations.
- CAPABLE Waitlist Control Group: Randomized to a wait-list control group to also receive the CAPABLE intervention after a specified waiting period.
Period: Overall Study
Arm/Group | Immediate CAPABLE | CAPABLE Waitlist Control Group
Started | 30 | 30
Completed (Of the 30 participants who completed the baseline assessment and were randomized to the immediate intervention group, 27 received the allocated intervention and completed the follow-up assessment. Three participants did not receive the allocated intervention because they were no longer interested (n=2) or died (n=1). All three of these subjects were withdrawn from the study prior to the start of the receipt of the intervention.) | 27 | 30
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CAPABLE Wait-list Control Group: Randomized to a wait-list control group to also receive the CAPABLE intervention after a specified waiting period.
- Total: Total of all reporting groups
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (6.8) | 62.7 (7.2) | 63.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 17 | 21 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 4 | 3 | 7
  Non-Hispanic Black | 19 | 12 | 31
  Asian, American Indian, or Alaska Native | 2 | 4 | 6
  Latino only | 0 | 2 | 2
  Biracial, multiracial, or multiethnic | 5 | 9 | 14
Education [Count of Participants; unit: Participants]
  Less than high school diploma | 6 | 12 | 18
  High school diploma or GED | 8 | 3 | 11
  Some college | 14 | 11 | 25
  Bachelor's degree or more | 2 | 4 | 6
Monthly Income [Mean (Standard Deviation); unit: US Dollars] — Average monthly income reported by participants in US Dollars.
  US Dollars | 924.98 (647.75) | 847.79 (480.47) | 884.36 (562.01)
Years living in current home [Mean (Standard Deviation); unit: Years] | 8.53 (7.55) | 7.20 (5.85) | 7.87 (6.73)
Years of homelessness [Mean (Standard Deviation); unit: years] | 6.15 (8.54) | 5.68 (6.51) | 5.91 (7.53)
Moderate or severe pain [Count of Participants; unit: Participants] — Assessed using an item from the 3-item PEG to assess average pain intensity (P), interference with enjoyment of life (E), and interference with general activity (G) on a 10-point Likert scale from 0 (no pain) to 10 (pain as bad as you can imagine). Moderate to severe pain was defined as any score greater than or equal to 4 on the 0 to 10 scale.
  Participants | 21 | 22 | 43
Three or more chronic health conditions [Count of Participants; unit: Participants] | 22 | 25 | 47
Falls in the past year [Mean (Standard Deviation); unit: Number of falls] | 7.17 (12.02) | 9.54 (20.46) | 8.47 (17.0)
Proportion of people with falls in past year [Mean (Standard Deviation); unit: Proportion of participants] | 0.67 (0.48) | 0.80 (0.41) | 0.73 (0.45)
Emergency room visits in past year [Mean (Standard Deviation); unit: Number of ER visits] | 2.10 (4.67) | 2.35 (3.57) | 2.22 (4.13)
Overnight hospitalizations in past year [Mean (Standard Deviation); unit: Number of hospitalizations] | 1.23 (2.87) | 0.97 (1.72) | 1.10 (2.36)

OUTCOME MEASURES:

1. Primary Outcome: Activities of Daily Living Limitations Score
Description: The modified Katz Activities of Daily Living (ADL) Index is an 8-item questionnaire that was completed by participants to rate their ability to perform daily activities, such as bathing, toileting, eating, and dressing, across a 5-point Likert scale (1 = no difficulty, 2 = a little difficulty, 3 = moderate difficulty, 4 = a lot of difficulty, 5 = unable to do). Items are summed to obtain a score with minimum and maximum values of 8 to 40, respectively, whereby higher scores represent greater difficulty performing ADLs.
Time Frame: Change of ability to perform activities of daily living from baseline to 6-month follow up (post-intervention).
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 27 | 30
Score on a scale
  Baseline | 17.07 [14.34 to 19.80] | 14.47 [12.58 to 16.35]
  Follow-up | 14.67 [12.63 to 16.70] | 13.17 [11.52 to 14.80]

2. Primary Outcome: Instrumental Activities of Daily Living Score
Description: The Brief Instrumental Functioning Scale will be used to assess ability to perform in six functions: bathing, dressing, going to toilet, transferring, continence, and feeding. Each area is assessed on a five point scale; participants rated their ability to perform daily tasks on a 5-point scale (1 = no difficulty, 2 = a little difficulty, 3 = moderate difficulty, 4 = a lot of difficulty, 5 = unable to do). Items are summed to obtain a score with minimum and maximum values of 8 to 40, respectively, whereby higher scores represent greater difficulty performing ADLs.
Time Frame: Change of ability to perform IADLs from baseline to 6-month follow up (post-intervention).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 27 | 30
score on a scale
  Baseline | 18.44 [15.09 to 21.80] | 15.07 [12.80 to 17.33]
  Follow-up | 15.96 [13.30 to 18.63] | 15.17 [12.82 to 17.50]

3. Primary Outcome: Depression
Description: Eight of the nine items in the Patient Health Questionnaire-9 were used to measure depression, rated on a 4-point scale of how frequently participants were bothered by the eight problems during a 2-week period (0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day). Items are summed to obtain a score with minimum and maximum values of 0 to 24, respectively, whereby higher scores represent greater depressive symptoms.
Time Frame: Change in depression symptoms from baseline to 6-month follow up (post-intervention).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 27 | 30
score on a scale
  Baseline | 11.78 [8.75 to 14.81] | 8.93 [6.11 to 11.75]
  Follow-up | 9.23 [7.49 to 10.98] | 9.47 [7.26 to 11.68]

4. Primary Outcome: Falls Efficacy
Description: Participants rated their confidence they could do each of 10 activities without falling on a 10-point scale, with total scores ranging from 10 (not very confident) to 100 (very confident) using the Tinetti Falls Efficacy Scale. Thus, higher scores indicate greater efficacy related to falls.
Time Frame: Change of falls efficacy from baseline to 6-month follow up (post-intervention).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 27 | 30
score on a scale
  Baseline | 64.59 [53.39 to 75.80] | 74.73 [66.16 to 83.31]
  Follow-up | 69.78 [60.47 to 79.09] | 73.80 [65.05 to 82.55]

5. Primary Outcome: Pain Interference With Usual Activities
Description: Pain interference with usual activities was assessed using an item from the 3-item PEG to assess average pain intensity (P), interference with enjoyment of life (E), and interference with general activity (G) on a 10-point Likert scale from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Change in the degree that pain interferes with usual activities from baseline to 6-month follow up (post-intervention).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 27 | 30
score on a scale
  Baseline | 6.26 [4.82 to 7.70] | 5.80 [4.54 to 7.06]
  Follow-up | 6.28 [5.04 to 7.53] | 5.44 [4.10 to 6.79]

6. Primary Outcome: Number of Falls in the Past Year or 6 Months
Description: Mean number of falls to the ground during the past year.
Time Frame: Number of falls in the past year reported at 6-month follow up.
Measure: Mean (95% Confidence Interval); unit: Number of falls
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 27 | 29
Number of falls | 1.22 [0.35 to 2.10] | 2.67 [1.06 to 4.28]

7. Secondary Outcome: Self-rated Health
Description: Self-rated health was measured on a 5-point scale (1 = excellent, 2 = very good, 3 = good, 4 = fair, 5 = poor). A higher score indicates poorer self-rated quality of health.
Time Frame: Change in self-rated health from baseline to 6-month follow up (post-intervention).
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 27 | 30
Score on a scale
  Baseline | 3.44 [2.99 to 3.90] | 3.97 [3.65 to 4.28]
  Follow-up | 3.44 [2.99 to 3.90] | 3.67 [3.31 to 4.02]

8. Secondary Outcome: Overall Quality of Life
Description: Quality of life was assessed using a single item: "Overall, how would you rate your quality of life?" Response options ranged from 1 = worst possible quality of life to 11 = best possible quality of life. Thus, a higher value indicated greater self-rated quality of life.
Time Frame: Change in quality of life from baseline to 6-month follow up (post-intervention).
Population: Analytic sample consisted of participants with valid information on the item(s) (e.g., who are not missing on item(s)). Two participants in the control group were excluded due to invalid responses.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 27 | 28
score on a scale
  Baseline | 6.48 [5.21 to 7.75] | 7.71 [6.32 to 9.09]
  Follow-up | 6.46 [5.42 to 7.51] | 6.68 [5.52 to 7.84]

9. Other Pre Specified Outcome: Proportion of Participants With Emergency Room Visits in Past 6 Months
Description: History of emergency room visits during the past year assessed by asking: "How many times did you visit the emergency room in the past year (since the last survey)?
Time Frame: Proportion of participants with ER visits in past 6 months reported at 6-month follow up.
Population: Analytic sample consisted of participants with valid information on the item(s) (e.g., who are not missing on item(s)). One participant in the treatment group and one participant in the control group were excluded due to invalid responses.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 26 | 29
Participants | 9 | 10

10. Other Pre Specified Outcome: Number of Emergency Room Visits in Past 6 Months
Description: History of emergency room visits during the past year assessed by asking: "How many times did you visit the emergency room in the past year (since the last survey)? Outcome is the mean number of ER visits in past 6 months.
Time Frame: Number of ER visits in past 6 months reported at follow up.
Population: as for outcome 9
Measure: Mean (90% Confidence Interval); unit: Number of ER visits
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 26 | 29
Number of ER visits | 0.85 [0.18 to 1.51] | 0.90 [0.19 to 1.60]

11. Other Pre Specified Outcome: Proportion of Participants With Hospitalizations in Past 6 Months
Description: History of hospitalization during the past year assessed by asking: How many times did you stay overnight in a hospital in the past year (since the last survey)?"
Time Frame: Proportion of participants with hospitalizations in past 6 months reported at 6-month follow-up
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 26 | 29
Participants | 6 | 6

12. Other Pre Specified Outcome: Number of Overnight Hospitalizations in Past 6 Months
Description: History of hospitalization during the past year assessed by asking: How many times did you stay overnight in a hospital in the past year (since the last survey)?" Outcome measure is the mean number of overnight hospitalizations in past 6 months.
Time Frame: Number of overnight hospitalizations in past 6 months reported at 6-month follow up.
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: Number of hospitalizations
Arm/Group | Immediate CAPABLE | CAPABLE Wait-list Control Group
Number analyzed (Participants) | 26 | 29
Number of hospitalizations | 1.77 [-0.66 to 4.19] | 0.31 [0.06 to 0.56]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the study time period from December 2020 through September 2021. Data on adverse events for each participant were collected during the 6 month period while enrolled in the study.
Groups:
- Immediate CAPABLE: Community Aging in Place-Advancing Better Living for Elders: CAPABLE is a client-directed home-based intervention that consists of time-limited services from an occupational therapist, a nurse, and a handyman working collaboratively with the older adult client. In most cases, the OT makes 6 visits, the RN makes 4 visits, and a handyman makes 1 to 2 visits to make any modifications to a person's home during a 6-month period. The first visits for the OT and RN are usually 90 minutes each and the later ones are usually an hour each. Visits are spaced to enable older adults to practice new strategies learned in the previous visit. There should be a clear "conclusion/graduation," with the older adult understanding how to use their new skills and apply them to future situations.
- CAPABLE Waitlist Control Group: Randomized to a waitlist control group to also receive the CAPABLE intervention after a specified waiting period.
Arm/Group | Immediate CAPABLE | CAPABLE Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Pilot study resulting in a small number of individuals assigned to each study arm and potentially limiting the ability to detect significant differences. Further, because assessments were based solely on self-report, objective measurements on outcomes such as hospitalization and health care utilization require additional investigation. This would allow for the development of a comprehensive picture of the intervention's potential to positively affect health and behavior outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT04076319/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT04076319/ICF_001.pdf